CLINICAL TRIAL: NCT02241837
Title: PARACHUTE III: A Multinational Trial to Evaluate the Longterm Safety of the Parachute System
Brief Title: PARACHUTE III Pressure Volume Loop Sub-Study
Acronym: PIII PV Loop
Status: Terminated | Type: Observational
Sponsor: CardioKinetix, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RD1051.B.3
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: heart failure; percutaneous; interventional cardiology; apical remodeling; LV dilatation; akinesis; dyskinesis; myocardial infarction
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Dyskinesias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective is to assess the longterm safety of the CardioKinetix Parachute Implant and Delivery System in the partitioning of the left ventricle in patients with heart failure due to ischemic heart disease. This sub-study has the additional assessment of improvement in Pressure Volume Loop and corresponding MSCT to allow improved monitoring of heart improvement after therapy. The PV Loop Substudy studies he effects of the Parachute Implant on pressure and volume as functional parameters of the Left Ventricle.

DETAILED DESCRIPTION:
While current therapies for heart failure (including but not limited to: medical management, cardiac resynchronization and ICDs) may represent the best treatment available today for the majority of HF patients, the medical community recognizes that pharmacologic therapy has been optimized to nearly the extent that is possible, and that any incremental improvements in the management of HF patients will now come from device based therapies. With this background, CardioKinetix has developed a catheter-based intravascular approach to ventricular partitioning using an implantable device. The purpose of this study is to assess the longterm safety of using the CardioKinetix Parachute device to isolate the malfunctioning portion of the left ventricle in patients with symptoms of HF due to ischemic heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study must meet ALL of the following inclusion criteria:

  1. Akinesis or dyskinesis due to myocardial infarction limited to anteroapical region
  2. Subject is not hospitalized at time of enrollment.
  3. NYHA Class at time of enrollment, either:

     * NYHA Class III or Ambulatory IV - if predominant during the 3-month period prior to enrollment
     * NYHA Class II - if diagnosed with NYHA Class III or IV during 3-month period prior to enrollment
  4. LVEF >15 or% and ≤ 40% as measured by echocardiography.
  5. Post LV MI structural heart dysfunction represented by LV wall motion abnormality (WMA) by echocardiography.
  6. Eligible for cardiac surgery
  7. Between 18 and 79 years of age (inclusive)
  8. Receiving appropriate medical treatment for heart failure according to the ACC/AHA 2009 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult during the three months prior to enrollment
  9. Provide written informed consent
  10. Agree to the protocol-required follow-up

Exclusion Criteria:

Candidates will be excluded from the study if ANY of the following conditions apply:

1. Untreated clinically significant coronary artery disease requiring intervention.
2. Acute MI (see MI definition) within 60 days of enrollment or patients with suspected evolving MI at time of enrollment
3. Cardiogenic shock within 72 hours of enrollment
4. Revascularization procedure (PCI or CABG) within 60 days of enrollment
5. Patient has received a pacemaker, ICD, or CRT device within 60 days of enrollment
6. History of aborted sudden cardiac death, if patient has not received an ICD and has potentially lethal ventricular arrhythmia, VT or VF
7. A known hypersensitivity or contraindication to aspirin, heparin, warfarin, nitinol (titanium and nickel alloy), or sensitivity to contrast media, which cannot be adequately pre medicated.
8. Aortic valve replacement or repair
9. Blood dyscrasia, history of bleeding diathesis or coagulopathy, or hypercoagulable states.
10. Active peptic ulcer or GI bleeding within the past 3 months
11. Patient has suffered a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months
12. History of Kawasaki's disease
13. Patient on dialysis or expected to require hemodialysis within 12 months
14. Patient has chronic liver disease
15. Impaired renal function that places patient at risk of contrast induced renal failure
16. Ongoing sepsis, including active endocarditis.
17. Co-morbidities associated with a life expectancy of less than 12-months or there are factors making echo and clinical follow-up difficult (no permanent address, etc.)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be open to all individuals who meet the inclusion/exclusion criteria. This is a prospective, multi-center, non-randomized trial.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Assessment of long term safety of the Parachute system from baseline to 1 year and annually | 5 years
  Assessment of long term safety as measured by site-reported device related MACE in real in real-world use of the Parachute Implant through 5 years of clinical follow-up.

SECONDARY OUTCOMES:
Change in Left Ventricular Volume Indices between baseline, 6 months, and annually | 6 months and annually to 5 years
  Change in Left Ventricular Volume Indexes (End Systolic {LVESVI} and End Diastolic {LVEDVI}) as measured by echocardiography from baseline to 6 months and annually to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Simon Redwood, MD, Principal Investigator — St. Thomas' Hospital
Locations (3):
- OLV Hospital Aalst, Aalst, Belgium
- Ferrarotto University Hospital Catania, Catania, Italy
- St. Thomas' Hospital, London, United Kingdom